CLINICAL TRIAL: NCT01711190
Title: The Effect of Trabeculectomy on Astigmatism.
Brief Title: Astigmatism Post-trabeculectomy
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Heleen Delbeke, MD, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S53708
Record Dates: First submitted 2012-02-24; First posted 2012-10-22 (Estimated); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Glaucoma
Keywords: glaucoma; trabeculectomy; astigmatism; intraocular pressure
MeSH Terms: conditions — Glaucoma; Astigmatism | interventions — Trabeculectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: trabeculectomy — Filtering surgery to reduce the intra-ocular pressure.

SUMMARY:
The aim of this project:

1. Confirming the modification in corneal astigmatism after trabeculectomy with MMC and intracameral administration of bevacizumab.
2. Medium-term follow up (6 months) of the induced corneal astigmatism.
3. Investigating correlations between postoperative astigmatism, particularly with the postoperative IOP.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma
* Normal tension glaucoma
* Pseudoexfoliation glaucoma
* Pigment dispersion glaucoma

Exclusion Criteria:

* Patients who refuse to sign the informed consent.
* Patients with primary angle closure glaucoma (PACG).
* Patients younger than 18 years old.
* Other ocular diseases besides glaucoma.
* Significant corneal opacities.
* Refractive error more than + or -6.00 diopters.
* Visual acuity less than 0.05
* Previous intra-ocular surgery (except cataract surgery more than six months preceding the trabeculectomy).
* Laser treatment for glaucoma within 6 months of the surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients having a primary trabeculectomy between January and April 2012 for glaucoma that was not adequately controlled with maximal tolerated medical therapy and/or laser therapy.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in ocular cylinder and axis untill 6 months after trabeculectomy. | pre-operative until 6 months post-operative
  Comparing the change in corneal cylinder, axis and IOP before the operation and 1,3 and 6 months after the operation. We will compare these vectors by vector analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Heleen Delbeke, MD, Principal Investigator — UZ Leuven
Locations (1):
- Sint-Raphaël hospital, Leuven, Vlaams-Brabant, Belgium